CLINICAL TRIAL: NCT02201186
Title: To Determine the Effect of Honey Enema in the Treatment of Patients With Acute Pouchitis (Pilot Study)
Brief Title: To Determine the Effect of Honey Enema in the Treatment of Patients With Acute Pouchitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Carl J Brown (Other)
Collaborators: Canadian Association of General Surgeons (Other)
Responsible Party: Sponsor-Investigator, Dr. Carl J Brown, Head, Division of General Surgery, clinical assistant professor of surgery at University of British Columbia, St. Paul's Hospital, Canada
Organization: St. Paul's Hospital, Canada (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H13-02740
Record Dates: First submitted 2014-07-19; First posted 2014-07-25 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Pouchitis
Keywords: honey enema for pouchitis
MeSH Terms: conditions — Pouchitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- manuka honey enema treatment (Experimental): Study patients diagnosed with acute pouchitis after bowel surgery for ulcerative colitis will perform manuka honey enemas twice a day for 30 days.
  Interventions: Other: Manuka honey enema

INTERVENTIONS:
Other: Manuka honey enema — Study patients diagnosed with acute pouchitis will perform manuka honey enemas twice a day for 30 days.

SUMMARY:
Patients with a bowel condition called ulcerative colitis have bowel surgery in which a portion of their bowel is removed and the reconnected at the small bowel to the anus. Sometimes, after the surgery, this connection part, the pouch, would be inflamed in a condition called Acute Pouchitis. Physicians usually treat them by prescribing antibiotics; however, some patients do not respond and need additional surgery. In this study, we will test an alternative treatment for this complication by performing manuka honey enemas twice a day for 30 days. This is a pilot study and ten patients will undergo enema treatment.

DETAILED DESCRIPTION:
Pouchitis is the most common long-term complication of ileal pouch-anal anastomosis (IPAA) in ulcerative colitis (UC). Pouchitis is defined as a clinical syndrome of watery, frequent, at times bloody stool accompanied by urgency, incontinence, abdominal cramps, malaise, and fever. The PDAI (Pouchitis Disease Activity Index) provides a standardized definition of pouchitis based on clinical, endoscopic, and histological markers. Pouchitis is defined as a score ≥ 7 and remission as a score < 7. Recently, the modified Pouchitis Disease Activity Index has been used to omit biopsy and histology from the standard PDAI. Omission of endoscopic biopsy and histology from the PDAI simplifies pouchitis diagnostic criteria, reduces the cost of diagnosis, and avoids delay associated with determining histology score, while providing equivalent sensitivity and specificity. Patients with acute pouchitis are managed routinely by antibiotics such as Ciprofloxacin and Metronidazole. This treatment has some side effects, is expensive, and fails to respond in some patients. Some patients who are unresponsive to antibiotic therapy will need to have a pouchectomy and ileostomy done.

On the other hand, multiple studies have shown that honey, especially manuka honey has anti-inflammatory, anti-bacterial, wound healing, and anti-ulcerous effects. Phenolic compounds in honey, such as flavonoids, have been reported to exhibit a wide range of biological activities, including antibacterial, antiviral, anti-inflammatory, antioxidant, antitumor, anti-allergic, and vasodilatory actions. This honey can clear infection, remove malodour, reduce inflammation and pain, cause edema and exudation to subside, and increase the rate of healing by stimulation of angiogenesis, granulation and epithelialization.

Due to problems associated with antibiotic therapy, such as side effects, cost and failure of some patients to respond, we are looking to find an alternative method for treating acute pouchitis. This study is designed to determine the effect of manuka honey on symptoms, signs and pathology of acute pouchitis patients. We will select patients with any of the signs and symptoms of pouchitis, such as abdominal pain, fever, frequency or urgency of defecation. Proctoscopy will be done before and after honey enema and the modified PDAI scores will be determined. The manuka honey enema will be administered twice a day, for one month. Then, the modified PDAI scores before and after completion of honey enema treatment of these patients, will be compared.

We know that bacterial overgrowth, ischemia, faecal stasis, recurrence of ulcerative colitis in the pouch, or possibly a novel third form of inflammatory bowel disease, are possible etiologies of pouchitis. We also know that manuka honey has anti-inflammatory and anti-bacterial properties. Some studies demonstrate that honey is effective in the treatment of induced colitis in animal models. However, there is no current literature on the effect of honey on colitis or pouchitis in humans. Based on the aforementioned properties of honey, and considering the probable etiologies of pouchitis, we expect that these patients will respond to this method of treatment.

Some research has been done on the effect of honey in the treatment of colitis in animal models, but there have been no clinical studies that have assessed this treatment in pouchitis, or even colitis, in humans. Considering the etiologies of pouchitis, such as inflammation and bacterial overgrowth, and considering the main effects of honey, such as anti-bacterial and anti-inflammatory efficacy, honey enema may be useful in the treatment of pouchitis. Our study is trying to determine the effect of manuka honey enema in the treatment of acute pouchitis. We will try to determine whether the honey enema helps to decrease inflammation and infection in the pouch, and thereby provide us with a safe alternative method for the treatment of pouchitis.

In this pilot study, we will select patients who have any of the signs and symptoms of acute pouchitis, such as abdominal pain, fever, frequency, or urgency of defecation. Proctoscopy will be performed on these patients. Ten patients with modified PDAI score ≥ 7 will receive honey enemas twice a day for one month. We chose a twice daily enema regimen, because patients with inflammatory bowel disease usually receive their enemas twice a day. We expect one month to be enough time, because the duration of antibiotic therapy for patients with acute pouchitis is about one month. Then, the PDAI score of these patients, before and after honey enema will be compared.

ELIGIBILITY:
Inclusion Criteria:

* have given written informed consent
* have been diagnosed with ulcerative colitis
* have had total colectomy and ileal pouch anal anastomosis before
* have presented with signs and symptoms of pouchitis within the last two months of signing the informed consent
* PDAI of greater than or equal to 7

Exclusion Criteria:

* patients who are unable to perform enema by themselves
* patients with an allergy to honey

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
PDAI score | within 2 weeks after the 30-day treatment
  PDAI score is a criterion for defining pouchitis. A PDAI score will be calculated from a proctoscopy assessment before treatment. Within two weeks after the treatment, another proctoscopy will be performed to determine the post-treatment PDAI score to see if there is a decrease in PDAI score for the study patients.

SECONDARY OUTCOMES:
Composite complications | throughout the 30-day honey enema treatment and within two weeks of the treatment completion date
  includes stool frequency (no different, 1-2 stools/day > postoperative usual, 3 or more stools/day > postoperative usual), rectal bleeding (none or rare or present daily), fecal urgency or abdominal cramps (none, occasional or usual), presence of fever (temperature >37.8° C), abdominal pain (no, occasional or usual) and readmission to hospital for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Brown, Principal Investigator — Saint Paul's Hospital
Locations (1):
- Saint Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Sandborn WJ, Tremaine WJ, Batts KP, Pemberton JH, Phillips SF. Pouchitis after ileal pouch-anal anastomosis: a Pouchitis Disease Activity Index. Mayo Clin Proc. 1994 May;69(5):409-15. doi: 10.1016/s0025-6196(12)61634-6. PMID 8170189
- [Background] Shen B, Achkar JP, Connor JT, Ormsby AH, Remzi FH, Bevins CL, Brzezinski A, Bambrick ML, Fazio VW, Lashner BA. Modified pouchitis disease activity index: a simplified approach to the diagnosis of pouchitis. Dis Colon Rectum. 2003 Jun;46(6):748-53. doi: 10.1007/s10350-004-6652-8. PMID 12794576
- [Background] Kafadar I, Moustafa F, Yalcin K, Klc BA. A rare adverse effect of metronidazole: nervous system symptoms. Pediatr Emerg Care. 2013 Jun;29(6):751-2. doi: 10.1097/PEC.0b013e318294f389. PMID 23736071
- [Background] Makhdoom A, Khan MS, Lagahari MA, Rahopoto MQ, Tahir SM, Siddiqui KA. Management of diabetic foot by natural honey. J Ayub Med Coll Abbottabad. 2009 Jan-Mar;21(1):103-5. PMID 20364754
- [Background] Kilicoglu B, Gencay C, Kismet K, Serin Kilicoglu S, Erguder I, Erel S, Sunay AE, Erdemli E, Durak I, Akkus MA. The ultrastructural research of liver in experimental obstructive jaundice and effect of honey. Am J Surg. 2008 Feb;195(2):249-56. doi: 10.1016/j.amjsurg.2007.04.011. PMID 18083132
- [Background] Cernak M, Majtanova N, Cernak A, Majtan J. Honey prophylaxis reduces the risk of endophthalmitis during perioperative period of eye surgery. Phytother Res. 2012 Apr;26(4):613-6. doi: 10.1002/ptr.3606. Epub 2011 Oct 6. PMID 22508360
- [Background] Hussein SZ, Mohd Yusoff K, Makpol S, Mohd Yusof YA. Gelam Honey Inhibits the Production of Proinflammatory, Mediators NO, PGE(2), TNF-alpha, and IL-6 in Carrageenan-Induced Acute Paw Edema in Rats. Evid Based Complement Alternat Med. 2012;2012:109636. doi: 10.1155/2012/109636. Epub 2012 Jul 1. PMID 22919407
- [Background] Medhi B, Prakash A, Avti PK, Saikia UN, Pandhi P, Khanduja KL. Effect of Manuka honey and sulfasalazine in combination to promote antioxidant defense system in experimentally induced ulcerative colitis model in rats. Indian J Exp Biol. 2008 Aug;46(8):583-90. PMID 18814487
- [Background] Viuda-Martos M, Ruiz-Navajas Y, Fernandez-Lopez J, Perez-Alvarez JA. Functional properties of honey, propolis, and royal jelly. J Food Sci. 2008 Nov;73(9):R117-24. doi: 10.1111/j.1750-3841.2008.00966.x. PMID 19021816